CLINICAL TRIAL: NCT04125108
Title: The Effect of a Pulmonary Rehabilitation on Lung Function and Exercise Capacity in Patients With Burn: a Prospective Randomized Single Blind Study
Brief Title: The Effect of a Pulmonary Rehabilitation on Lung Function and Exercise Capacity in Patients With Burn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hangang Sacred Heart Hospital (Other)
Collaborators: National Research Foundation of Korea (Other); Hallym University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HangangSHH-6
Record Dates: First submitted 2019-10-10; First posted 2019-10-14 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2019-10

CONDITIONS: Inhalation Injury; Pulmonary Disease
Keywords: burn; Pulmonary Function Test; Pulmonary Rehabilitation
MeSH Terms: conditions — Lung Diseases; Burns

STUDY DESIGN:
Intervention Model Description: The patients with inhalation injury, chest and neck burn injury were included. The burn surface area of chest and neck are more than 50% of the anterior or posterior trunk areas.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pulmonary rehabilitation group (Experimental): The experimental group was to participate in a 12-week pulmonary rehabilitation program supplemented with an individualized and supervised exercise-training program.
  Interventions: Other: pulmonary rehabilitation
- control group (No Intervention): The control group was to participate in a 12-week conventional rehabilitation program.

INTERVENTIONS:
Other: pulmonary rehabilitation — Pulmonary rehabilitation programs were designed to include both 30 minutes resistance and 30 minutes aerobic exercises. Eight basic resistnace exercises were used incorporating, bench press, leg press, leg curl, leg extension, toe raises, biceps curl, triceps curl, shoulder press. Additionally each exercise training session also included aerobic conditioning exercises ona treadmill or cycle ergometer. Aerobic exercise training was carried out 5 days per week, with each session lasting 30 minutes. All exercise sessions were preceded by a 5-minutes warm up period on a treadmill set.
  Arms: pulmonary rehabilitation group

SUMMARY:
Inhalation burn injury and lung complications caused by large surface burns occurring during a fire remains a serious problem. Pulmonary rehabilitation has been used successfully to improve pulmonary function(PF) in patients with chronic obstructive pulmonary disease. But there were no studies that pulmonary rehabilitation induce improvements in PF in patient with large surface burn and inhalation injury.

The investigators will performe pulmonary function and respiratory muscles strength evaluation in 40 patients with thermal injury in order to evaluate the effects of pulmonary rehabilitation in patients with thermally injury.

DETAILED DESCRIPTION:
The investigators will performe pulmonary function and respiratory muscles strength evaluation in 40 patients with thermal injury in order to evaluate the effects of pulmonary rehabilitation in patients with thermally injury.

The investigators will study 40 patients who had burn injury. Burned patients will be randomized into two groups. The experimental group(EG) will participate in a 12-week pulmonary rehabilitation program daily for 60 minutes. The control group(CG) will participate in a 12-week conventional exercise program daily for 60 minutes. Spirometer will be done to evaluate pulmonary function. Pulmonary function tests include forced vital capacity(FVC), 1 second forced expiratory volume(FEV1), forced expiratory flow rate between 25 and 75% of the FVC(FEF 25-75) FEV1/FVC ratio expressed as a percentage(FEV1/FVC %) and peak expiratory flow(PEF). Maximum voluntary ventilation(MVV) and respiratory muscles strength(MEP[maximal expiratory pressure], MIP[maximal inspiratory pressure]) will be measured by mouth pressure-meter in sitting position. Pulmonary function tests will be performed for all groups at baseline and after 12 weeks programs. A 6-minute walk test and health-related quality of life will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* inhalation injury
* The burn surface area of chest and neck are more than 50% of the anterior or posterior trunk areas.

Exclusion Criteria:

* vocal cord palsy
* who were intubated
* had a tracheostomy
* anoxic brain injury
* psychologicical disorders
* quadriplegia
* severe cognitive disorders
* who took medications that affect pulmonary function.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
FVC | 12 weeks
  forced vital capacity(%)
FEV1 | 12 weeks
  1 second forced expiratory volume(%)
FEV1/FVC ratio | 12 weeks
  FEV1/FVC ratio expressed as a percentage(%)

SECONDARY OUTCOMES:
MEP | 12 weeks
  maximal expiratory pressure
MIP | 12 weeks
  maximal inspiratory pressure
gait performance | 12 weeks
  6-minute walk test

CONTACTS AND LOCATIONS:
Locations (1):
- Hangang Sacred Heart Hospital, Seoul, Yeong-deungpo-Dong, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Al-Mousawi AM, Williams FN, Mlcak RP, Jeschke MG, Herndon DN, Suman OE. Effects of exercise training on resting energy expenditure and lean mass during pediatric burn rehabilitation. J Burn Care Res. 2010 May-Jun;31(3):400-8. doi: 10.1097/BCR.0b013e3181db5317. PMID 20354445
- [Result] Ring J, Heinelt M, Sharma S, Letourneau S, Jeschke MG. Oxandrolone in the Treatment of Burn Injuries: A Systematic Review and Meta-analysis. J Burn Care Res. 2020 Jan 30;41(1):190-199. doi: 10.1093/jbcr/irz155. PMID 31504621